CLINICAL TRIAL: NCT05049590
Title: Acute Normovolemic Hemodilution (ANH) in Complex Cardiac Surgery
Brief Title: Acute Normovolemic Hemodilution in Complex Cardiac Surgery
Acronym: ANH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-000469
Record Dates: First submitted 2021-06-22; First posted 2021-09-20 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Cardiac Surgery; Acute Kidney Injury; Congenital Heart Disease; Aortic Surgery
Keywords: acute normovolemic hemodilution; complex cardiac surgery; transfusions; acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury; Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Perform blood conservation in the operating room (OR).
  Interventions: Biological: Acute normovolemic hemodilution (ANH)
- Control Group (No Intervention): Blood conservation will not be performed in the OR.

INTERVENTIONS:
Biological: Acute normovolemic hemodilution (ANH) — A blood conservation technique that removes whole blood (~8-10cc/kg) from a patient in the operating room prior to incision.
  Arms: Intervention Group

SUMMARY:
Postoperative bleeding in cardiac surgery is a frequent complication, and cardiac surgery utilizes 15-20% of the national blood supply. Packed red blood cells (pRBCs) are associated with worse short and long term outcomes. For each unit transfused, there is an additive risk of mortality (death) and cardiac adverse events. Despite current guidelines and numerous approaches to bleeding reduction, >50% of the patients undergoing cardiac surgery receive transfusions. Acute normovolemic hemodilution (ANH), a blood conservation technique that removes whole blood from a patient immediately prior to surgery, could be a valuable method to reduce transfusion in complex cardiac surgery. At the University of California, Los Angeles (UCLA), ANH is routinely utilized in patients who refuse allogenic blood transfusions such as Jehovah's Witnesses. ANH has been shown to be safe with minimal risk to patients. ANH has been studied in simple cardiac surgery, such as coronary artery bypass grafting, however it has not been studied in complex cardiac surgery, such as aortic surgery and adult congenital heart disease. ANH has been demonstrated to reduce pRBC transfusion in lower risk cardiac surgery without any significant complications. Complex heart surgery utilizes more blood products. This study could identify the benefits of ANH in a higher risk surgical group.

DETAILED DESCRIPTION:
Adult patients undergoing complex heart surgery will be randomized to 1 of 2 groups using block randomization: the intervention arm receiving acute normovolemic hemodilution (ANH) or the control arm receiving standard of care.

As day of surgery hemoglobin (Hgb)/hematocrit (Hct) is critical to the final determination for study participation, patients will be randomized to control or intervention arms after the first intraoperative arterial blood gas (ABG) is obtained. The Hb/Hct obtained from this ABG is used to determine the postdilutional hematocrit using specific pre-ANH and post-ANH equations. Patients with pre-ANH or post-ANH postdilutional Hct lower than 22-24 will not be eligible for inclusion in the ANH arm of the study.

For the Study Group: Using sterile techniques, ANH is performed by removing 8-10cc/kg of whole blood with a maximum of 700cc, from the patient in the OR prior to incision. Whole blood will be collected and stored at room temperature. Hemodynamics are assessed during whole blood removal to ensure adequate stability. ANH will be discontinued if the patient becomes hemodynamically unstable (i.e. significant hypotension greater than 20% reduction from pre-ANH, unstable arrhythmia, evidence of myocardial ischemia or evidence of worsening myocardial function). After whole blood removal, the patient is hydrated to maintain isovolemia with an equivalent volume of crystalloid and/or colloid given, and the blood is stored in the OR at room temperature. After cardiopulmonary bypass (CPB) is complete, the whole blood is returned to the patient. Whole blood stored at room temperature will be transfused within 8 hours of initial collection. After 8 hours, ANH whole blood will be considered expired and will be transfused back to the patient prior to expiration and not discarded. Laboratory coagulation and ROTEM studies (assess blood clotting) will be resent after the ANH blood is returned to the patient. Transfusion requirement will be continuously reassessed based upon laboratory values and surgical assessment of clinical bleeding.

For the Control Group: Blood conservation will not be performed in the OR. Coagulation labs (i.e. platelet count, fibrinogen level and ROTEM studies) are sent while the patient in on bypass. After separation from bypass, coagulation laboratory studies and clinical bleeding are assessed in collaboration with the surgeon. Based on laboratory values and surgical assessment, allogenic transfusions (donor/recipient not the same person) occur in a targeted fashion (i.e. clinical bleeding with platelet count less than 150 x10E3/uL and a ROTEM results indicative of inadequate clot strength will result in platelet transfusion). Transfusion requirements are continuously reassessed based upon updated laboratory values and surgical assessment of clinical bleeding.

Data will also be collected and recorded from the medical record for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients presenting for elective cardiac surgery
* Surgical procedures to include:

  * Redo surgery
  * Adult congenital heart disease surgery (ACHD)
  * Aortic surgery including aortic surgery requiring deep hypothermic circulatory arrest

Exclusion Criteria:

* low risk cardiac surgery
* cardiac surgery not requiring cardiopulmonary bypass
* baseline anemia (Hgb < 13 for men and 12 for women)
* post-dilution Hct < 21-24 (basis for this is increased risk of AKI on CPB with Hct 21-22)
* preop treatment for anemia
* high-risk ischemia lesions (critical left main, multi-vessel disease, active/recent chest pain, unstable angina, presence of a balloon pump, recent history of myocardial infarction (MI) either non-ST elevation MI (NSTEMI) / ST-elevation MI (STEMI), regional wall motion abnormalities on echo)
* low left ventricular systolic function (LVEF < 35-40%) - decompensated heart failure
* Hypertrophic obstructive cardiomyopathy (HOCM) patients with significant left ventricular outflow tract (LVOT) gradients
* history of recent blood transfusion
* history of recent gastrointestinal (GI) bleed
* patient refusal to participate in the study
* severe aortic stenosis (AS) with reduced LVEF
* pulmonary hypertension
* underlying significant liver disease impairing synthetic function (elevated PT/INR or PTT) at baseline
* clotting disorders, inherited or acquired or iatrogenic coagulopathy (i.e. thrombocytopenia, pancytopenia)
* baseline chronic kidney disease (CKD) stage 3/above or End-stage renal disease (ESRD) +/- hemodialysis
* hemodynamically unstable patients including sepsis/recently treated sepsis
* preoperative extracorporeal membrane oxygenation (ECMO) or high suspicion for postoperative ECMO
* emergent cases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Packed red blood cells (pRBC) | 24 hours
  Total transfusion of pRBC units administered 24 hours post-operatively.
Packed red blood cells (pRBC) | 48 hours
  Total transfusion of pRBC units administered 48 hours post-operatively.
Packed red blood cells (pRBC) | 72 hours
  Total transfusion of pRBC units administered 72 hours post-operatively.

SECONDARY OUTCOMES:
Maximum Intraoperative Vasoactive-Inotropic Score | Conclusion of intraoperative procedure
  The maximum intraoperative vasoactive-inotropic score quantifies the amount of cardiovascular support required. The score is calculated based on the highest dose of vasoactive or inotropic drugs used after the conclusion of cardiopulmonary bypass during the intraoperative period. At our institution, the score range is between 0 and 125 with higher scores equating with higher need for support. The drugs included in the calculation include vasopressin, epinephrine, norepinephrine, levosimendan, olprinone, methylene blue, milrinone, phenylephrine, terlipressin, angiotensin II, dobutamine, dopamine and enoximone.
Maximum 24 Hour Vasoactive-Inotropic Score | 24 hours
  The maximum 24 hour vasoactive-inotropic score quantifies the amount of cardiovascular support required over the first 24 hours post-operatively. The score is calculated based on the highest doses of vasoactive and inotropic drugs used during the first 24 hour period postoperatively. At our institution, the score range is between 0 and 125 with higher scores equating with higher need for support. The drugs included in the calculation include vasopressin, epinephrine, norepinephrine, levosimendan, olprinone, methylene blue, milrinone, phenylephrine, terlipressin, angiotensin II, dobutamine, dopamine and enoximone.
Maximum 48 Hour Vasoactive-Inotropic Score | 48 hours
  The maximum 48 hour vasoactive-inotropic score quantifies the amount of cardiovascular support required over the first 48 hours post-operatively. The score is calculated based on the highest doses of vasoactive and inotropic drugs used during the first 48 hour period postoperatively. At our institution, the score range is between 0 and 125 with higher scores equating with higher need for support. The drugs included in the calculation include vasopressin, epinephrine, norepinephrine, levosimendan, olprinone, methylene blue, milrinone, phenylephrine, terlipressin, angiotensin II, dobutamine, dopamine and enoximone.
Maximum 72 Hour Vasoactive-Inotropic Score | 72 hours
  The maximum 72 hour vasoactive-inotropic score quantifies the amount of cardiovascular support required over the first 72 hours post-operatively. The score is calculated based on the highest doses of vasoactive and inotropic drugs used during the first 72 hour period postoperatively. At our institution, the score range is between 0 and 125 with higher scores equating with higher need for support. The drugs included in the calculation include vasopressin, epinephrine, norepinephrine, levosimendan, olprinone, methylene blue, milrinone, phenylephrine, terlipressin, angiotensin II, dobutamine, dopamine and enoximone.
Acute Kidney Injury (AKI) | 72 hours
  Incidence of AKI based on RIFLE (Risk, Injury, Failure, Loss of kidney function, and End-stage kidney disease)/KDIGO (Kidney Disease Improving Global Outcomes) criteria within first 72 hours post-op.
24 Hour Chest Tube Output | 24 Hours
  Chest tubes are placed by surgeons at the conclusion of the cases and attached to chest drains. The volume of chest tube drainage is recorded by nurses every 8 hours. The total volume of chest tube output collected in the chest drains will be calculated for the first 24 hours postoperatively.
48 Hour Chest Tube Output | 48 Hours
  Chest tubes are placed by surgeons at the conclusion of the cases and attached to chest drains. The volume of chest tube drainage is recorded by nurses every 8 hours. The total volume of chest tube output collected in the chest drains will be calculated for the first 48 hours postoperatively.
72 Hour Chest Tube Output | 72 Hours
  Chest tubes are placed by surgeons at the conclusion of the cases and attached to chest drains. The volume of chest tube drainage is recorded by nurses every 8 hours. The total volume of chest tube output collected in the chest drains will be calculated for the first 72 hours postoperatively.
24 Hour Prothrombin time (PT) | 24 hours
  The maximum and minimum prothrombin time (units: seconds) that is collected between hours 0 and 24 postoperatively will be reported.
48 Hour Prothrombin time (PT) | 48 hours
  The maximum and minimum prothrombin time (units: seconds) that is collected between hours 24 and 48 postoperatively will be reported.
72 Hour Prothrombin time (PT) | 72 hours
  The maximum and minimum prothrombin time (units: seconds) that is collected between hours 48 and 72 postoperatively will be reported.
24 Hour International Normalized Ratio (INR) | 24 hours
  The maximum and minimum international normalized ratio (units: N/A) that is collected between hours 0 and 24 postoperatively will be reported.
48 Hour International Normalized Ratio (INR) | 48 hours
  The maximum and minimum international normalized ratio (units: N/A) that is collected between hours 24 and 48 postoperatively will be reported.
72 Hour International Normalized Ratio (INR) | 72 hours
  The maximum and minimum international normalized ratio (units: N/A) that is collected between hours 48 and 72 postoperatively will be reported.
24 Hour Activated Partial Thromboplastin time (aPTT) | 24 hours
  The maximum and minimum activated partial thromboplastin time (units: seconds) that is collected between hours 0 and 24 postoperatively will be reported.
48 Hour Activated Partial Thromboplastin time (aPTT) | 48 hours
  The maximum and minimum activated partial thromboplastin time (units: seconds) that is collected between hours 24 and 48 postoperatively will be reported.
72 Hour Activated Partial Thromboplastin time (aPTT) | 72 hours
  The maximum and minimum activated partial thromboplastin time (units: seconds) that is collected between hours 48 and 72 postoperatively will be reported.
24 Hour Fibrinogen | 24 hours
  The maximum and minimum fibrinogen (units: mg/dL) that is collected between hours 0 and 24 postoperatively will be reported.
48 Hour Fibrinogen | 48 hours
  The maximum and minimum fibrinogen (units: mg/dL) that is collected between hours 24 and 48 postoperatively will be reported.
72 Hour Fibrinogen | 72 hours
  The maximum and minimum fibrinogen (units: mg/dL) that is collected between hours 48 and 72 postoperatively will be reported.
24 Hour Platelet Count | 24 hours
  The maximum and minimum platelet count (units: 10E3/uL) that is collected between hours 0 and 24 postoperatively will be reported.
48 Hour Platelet Count | 48 hours
  The maximum and minimum platelet count (units: 10E3/uL) that is collected between hours 24 and 48 postoperatively will be reported.
72 Hour Platelet Count | 72 hours
  The maximum and minimum platelet count (units: 10E3/uL) that is collected between hours 48 and 72 postoperatively will be reported.
24 Hour Hemoglobin (Hgb) | 24 hours
  The maximum and minimum hemoglobin (units: g/dL) that is collected between hours 0 and 24 postoperatively will be reported.
48 Hour Hemoglobin (Hgb) | 48 hours
  The maximum and minimum hemoglobin (units: g/dL) that is collected between hours 24 and 48 postoperatively will be reported.
72 Hour Hemoglobin (Hgb) | 72 hours
  The maximum and minimum hemoglobin (units: g/dL) that is collected between hours 48 and 72 postoperatively will be reported.
24 Hour Hematocrit (Hct) | 24 hours
  The maximum and minimum hematocrit (units: %) that is collected between hours 0 and 24 postoperatively will be reported.
48 Hour Hematocrit (Hct) | 48 hours
  The maximum and minimum hematocrit (units: %) that is collected between hours 24 and 48 postoperatively will be reported.
72 Hour Hematocrit (Hct) | 72 hours
  The maximum and minimum hematocrit (units: %) that is collected between hours 48 and 72 postoperatively will be reported.
Rotational Thromboelastometry FIBTEM Maximum Clot Firmness (FIBTEM MCF) | During intraoperative period
  While on cardiopulmonary bypass, rotational thromboelastometry, a point of care viscoelastic test of hemostasis in whole blood, is completed which allows for the quantitative assessment of global clot formation, strength and dissolution. The FIBTEM assesses clot formation via the extrinsic pathway in the presence of cytochalasin D with the resulting clot dependent upon only fibrin formation and fibrin polymerization. The FIBTEM maximum clot firmness (units: mm) is the greatest vertical amplitude of the trace and is indicative of the absolute strength of the clot due to fibrin. A low MCF, less than 7mm, is suggestive of decreased fibrinogen level or polymerization.
Rotational Thromboelastometry HEPTEM/EXTEM Maximum Clot Firmness (HEPTEM/EXTEM MCF) | During intraoperative period
  While on cardiopulmonary bypass, rotational thromboelastometry, a point of care viscoelastic test of hemostasis in whole blood, is completed which allows for the quantitative assessment of global clot formation, strength and dissolution. The HEPTEM assesses clot formation via the intrinsic pathway in the presence of heparinase thereby inactivating circulating heparin, which is appropriate during cardiopulmonary bypass when the patient is systematically heparinized. The EXTEM assesses clot formation via the extrinsic pathway. The HEPTEM/EXTEM maximum clot firmness (units: mm) is the greatest vertical amplitude of the trace and is indicative of the absolute strength of the clot due to fibrinogen and platelets. A low MCF, less than 50mm, is suggestive of decreased platelet number/function or decreased fibrinogen level or polymerization.
Rotational Thromboelastometry EXTEM Clotting Time (EXTEM CT) | During intraoperative period
  While on cardiopulmonary bypass, rotational thromboelastometry, a point of care viscoelastic test of hemostasis in whole blood, is completed which allows for the quantitative assessment of global clot formation, strength and dissolution. The EXTEM assesses clot formation via the extrinsic pathway. The EXTEM clotting time (units: seconds) is the time from start of the measurement until initiation of clotting and is indicative of coagulation factor quantity and function. A high CT, greater than 80 seconds, is suggestive of inadequate clotting factors.
Rotational Thromboelastometry EXTEM Clotting Time (EXTEM A20) | During intraoperative period
  While on cardiopulmonary bypass, rotational thromboelastometry, a point of care viscoelastic test of hemostasis in whole blood, is completed which allows for the quantitative assessment of global clot formation, strength and dissolution. The EXTEM assesses clot formation via the extrinsic pathway. The EXTEM clotting time (units: seconds) is the time from start of the measurement until initiation of clotting and is indicative of coagulation factor quantity and function. A high CT, greater than 80 seconds, is suggestive of inadequate clotting factors.
Rotational Thromboelastometry HEPTEM Clotting Time (HEPTEM CT) | During intraoperative period
  While on cardiopulmonary bypass, rotational thromboelastometry, a point of care viscoelastic test of hemostasis in whole blood, is completed which allows for the quantitative assessment of global clot formation, strength and dissolution. The HEPTEM assesses clot formation via the intrinsic pathway in the presence of heparinase thereby inactivating circulating heparin, which is appropriate during cardiopulmonary bypass when the patient is systematically heparinized. The HEPTEM clotting time (units: seconds) is the time from start of the measurement until initiation of clotting and is indicative of coagulation factor quantity and function. A high HEPTEM CT, greater than 200 seconds, is suggestive of inadequate clotting factors.
Post-cardiopulmonary bypass HEPTEM/EXTEM MCF | In the operating room (OR) during surgery.
  We will assess the pre- and post-ANH ROTEM to determine for hemostasis quality by analyzing the viscoelastic properties of the patient's blood clot. We will compare the baseline ROTEM to the on-bypass and post-ANH ROTEM.
Cerebral oximetry using near infrared spectroscopy derived tissue oxygenation as a marker of perfusion | In the OR during surgery.
  Intraoperatively, cerebral oximetry using near infrared spectroscopy (NIRS)derived tissue oxygenation is used to grossly monitor grossly cerebral perfusion of the left and right cerebral hemispheres. Values are reported on a scale of 0 (lowest) to 100 (highest). A baseline cerebral oximetry is obtained upon application of the monitoring stickers. Throughout the case, the left and right cerebral oximetry values are reported. We will compare the change in cerebral oximetric value from baseline to values at bypass initiation, bypass separation, after ANH administration and at the case conclusion.
Change in mixed venous oxygen saturation as a marker of perfusion | 72 hours
  Using a continuous oximetry pulmonary artery catheter, intraoperative and postoperative mixed venous oxygen saturations will be recorded. We will compare the baseline mixed venous oxygen saturation obtained after PAC to the mixed venous oxygen saturation at bypass initiation, bypass separation, post-ANH administration, case conclusion, upon ICU arrival and then 24, 48, 72 hours post-op (or until the PAC is discontinued or discharge from the ICU). A subset of patients may not have PAC placed due to the nature of the surgery. We will not trend/monitor mixed venous in those patients.
Perfusion markers (lactate) | 72 hours
  Intra-op and post-op lactate values. We will compare the baseline lactate (from pre-induction/induction ABG) to the lactate at bypass initiation (30 mins after bypass initiation), at bypass separation, post-ANH administration, case conclusion, upon ICU arrival and then 24/48/72 hours post-op or until discharge from the ICU.
Delirium | Two times per day for up 72 hours post-op or until discharge from the ICU, whichever came first
  Confusion Assessment Method for the ICU (CAM-ICU)
Number of patients with infection/sepsis | 72 hours post-op or until discharge from the ICU, whichever came first
  ICU nurses complete a postoperative severe sepsis/shock screen based on white cell counts, temperature, hemodynamics (heart rate and blood pressure) and the presence of any known infectious source (i.e. positive urine culture, blood culture, etc). The total number of patients in the treatment and control arms with reported positive severe sepsis/shock screen will be recorded.
Mortality | An average of 5-10 days until discharge from the hospital, whichever came first
  In-hospital mortality
Platelets (PLT) | 24 hours
  Total transfusion of PLT units administered 24 hours post-operatively.
Platelets (PLT) | 48 hours
  Total transfusion of PLT units administered 48 hours post-operatively.
Platelets (PLT) | 72 hours
  Total transfusion of PLT units administered 72 hours post-operatively.
Fresh frozen plasma (FFP) | 24 hours
  Total transfusion of FFP units administered 24 hours post-operatively.
Fresh frozen plasma (FFP) | 48 hours
  Total transfusion of FFP units administered 48 hours post-operatively.
Fresh frozen plasma (FFP) | 72 hours
  Total transfusion of FFP units administered 72 hours post-operatively.
Cryoprecipitate (cryo) | 24 hours
  Total transfusion of cryo units administered 24 hours post-operatively.
Cryoprecipitate (cryo) | 48 hours
  Total transfusion of cryo units administered 48 hours post-operatively.
Cryoprecipitate (cryo) | 72 hours
  Total transfusion of cryo units administered 72 hours post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Lorraine Lubin, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Ronald Reagan UCLA Medical Center, Department of Anesthesiology & Perioperative Medicine, Los Angeles, California, United States

REFERENCES:
- [Background] Barile L, Fominskiy E, Di Tomasso N, Alpizar Castro LE, Landoni G, De Luca M, Bignami E, Sala A, Zangrillo A, Monaco F. Acute Normovolemic Hemodilution Reduces Allogeneic Red Blood Cell Transfusion in Cardiac Surgery: A Systematic Review and Meta-analysis of Randomized Trials. Anesth Analg. 2017 Mar;124(3):743-752. doi: 10.1213/ANE.0000000000001609. PMID 27669554
- [Background] Zhou ZF, Jia XP, Sun K, Zhang FJ, Yu LN, Xing T, Yan M. Mild volume acute normovolemic hemodilution is associated with lower intraoperative transfusion and postoperative pulmonary infection in patients undergoing cardiac surgery -- a retrospective, propensity matching study. BMC Anesthesiol. 2017 Jan 26;17(1):13. doi: 10.1186/s12871-017-0305-7. PMID 28122491